CLINICAL TRIAL: NCT05683145
Title: University of Colorado - Restoring Efficient Sleep After TBI (CU-REST)
Brief Title: University of Colorado - Restoring Efficient Sleep After TBI
Acronym: CU-REST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: Colorado Traumatic Brain Injury Trust Fund (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMIRB 22-1169
Record Dates: First submitted 2022-12-14; First posted 2023-01-12 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Insomnia; Traumatic Brain Injury
Keywords: computerized intervention; insomnia; traumatic brain injury; clinician guided
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: parallel, two-arm, randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized Cognitive Behavioral Therapy for Insomnia (Experimental): Self-guided computerized CBT-I program with assistance from a licensed mental health professional.
  Interventions: Behavioral: Computerized Cognitive Behavioral Therapy for Insomnia
- Enhanced Treatment as Usual (No Intervention): ETU is defined as treatment per usual which is enhanced by participating in data collection related to study participation.

INTERVENTIONS:
Behavioral: Computerized Cognitive Behavioral Therapy for Insomnia — This is a computerized version of cognitive behavioral therapy for insomnia that is augmented by support from a licensed mental health professional. The intervention consists of 6 modules designed to provide education regarding sleep and insomnia, establish behavioral modifications to reduce insomnia symptoms, and monitor progress. Participants will be able to complete these intervention at their own pace, which will take between 6-9 weeks.
  Arms: Computerized Cognitive Behavioral Therapy for Insomnia

SUMMARY:
Sleep disturbance is a common condition following traumatic brain injury (TBI) and impairs recovery and quality of life. While efficacious interventions exist many are not accessible to all patients due to a variety of factors (e.g., rurality, access to providers). Further, many of the available treatments have not been validated for individuals with moderate/severe TBI. The proposed study will evaluate a guided computerized version of cognitive behavioral therapy for insomnia (cCBT-I) against enhanced treatment as usual (ETU) in individuals with moderate/severe TBI.

DETAILED DESCRIPTION:
Individuals with a history of moderate to severe TBI experience multi-faceted sleep problems, including greater daytime sleepiness, lesser total sleep time, and difficulties with initiating, maintaining, and self-monitoring sleep. Such sleep complaints may reflect underlying sleep conditions such as insomnia, the prevalence of which is significantly greater among individuals with TBI (29%) compared to members of the general population (10%). As such, treatment of insomnia among individuals with moderate to severe TBI is expected to produce wide-ranging benefits in regards to short- and long-term rehabilitation. Among members of the general population, cognitive behavioral therapy for insomnia (CBT-I) is considered the gold standard for treating insomnia. CBT-I focuses on improving sleep quality via cognitive therapy, behavioral techniques, and psychoeducation. However, access to in-person treatment has been limited by cost, insufficient numbers of adequately trained healthcare providers, and patient perceptions regarding the efficacy of the intervention, as well as additional barriers that may be particularly pertinent for those living with moderate to severe TBI (e.g., limited transportation). Optimally, an intervention for those with TBI and insomnia would show efficacy at reversing sleep inefficiency, and be able to be used with minimal stigma. In addition, the intervention should be highly accessible, low cost, self-sustaining (e.g., portable), and with minimal side effects.

Computerized versions of CBT-I assist in reducing barriers to access and have been found to be acceptable and efficacious in a variety of populations, including those with mild TBI. To date, research among those with moderate to severe TBI has been limited. This study will address this gap by examining the efficacy of a guided computerized CBT-I (CCBT-I) intervention for those with moderate to severe TBI and insomnia. That is, we will implement a free, computerized version of CBT-I, provided in conjunction with guidance (e.g., prompts or reminders to complete modules, help or support using the program and/or completing the modules) by a licensed mental health professional (Study Clinician). As participants will be recruited from the community at-large across the State of Colorado, it is believed that findings will be highly generalizable.

Moreover, both geography (where an individual resides) and challenges with transportation create barriers to treatment access and research participation among those living with moderate to severe TBI. As such, all study procedures will be completed remotely. During the Coronavirus Disease 2019 (COVID-19) pandemic, members of this study team explored and implemented multiple methods to facilitate remote research participation (e.g., video conferencing, data collection via Research Electronic Data Capture [REDCap], mailing study data collection devices). Employing such methods will allow individuals in both rural and urban areas across Colorado to participate.

ELIGIBILITY:
Inclusion Criteria:

* History of post-acute (i.e., at least one year after injury) moderate to severe traumatic brain injury
* Current insomnia
* Reliable access to the internet
* Ability to provide informed consent

Exclusion Criteria:

* Active substance dependence, excluding cannabis
* Current psychosis
* Bipolar disorder
* Current sleep disorders other than insomnia, including sleep apnea
* Irregular work schedule, shift work, and/or life changes (e.g., newborn) interfering with regular sleep patterns.
* Currently receiving psychological treatment for insomnia
* Pregnancy
* Currently involved in another research interventional trial targeting insomnia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Change from baseline to post-intervention (CCBT-I arm) or 9 weeks following randomization (ETU arm).
  The change in the total score of the ISI, compared across study arms, will be used as the outcome.

OTHER OUTCOMES:
Total sleep time - discrepancy between sleep diary and actigraphy | Two timepoints: One week prior to the start of the intervention and for the week immediately following completion of the intervention
  Change in the discrepancy between sleep diary- and actigraphy-derived total sleep time will be evaluated for the CCBT-I arm.
Sleep onset latency - discrepancy between sleep diary and actigraphy | Two collection periods: One week prior to the start of the intervention and for the week immediately following completion of the intervention
  Change in the discrepancy between sleep diary- and actigraphy-derived sleep onset latency will be evaluated for the CCBT-I arm.
Wake after sleep onset - discrepancy between sleep diary and actigraphy | Two collection periods: One week prior to the start of the intervention and for the week immediately following completion of the intervention
  Change in the discrepancy between sleep diary- and actigraphy-derived wake after sleep onset will be evaluated for the CCBT-I arm.
Sleep efficiency - discrepancy between sleep diary and actigraphy | Two collection periods: One week prior to the start of the intervention and for the week immediately following completion of the intervention
  Change in the discrepancy between sleep diary- and actigraphy-derived sleep efficiency will be evaluated for the CCBT-I arm.
Nature and duration of guidance needed to compete intervention | Through study completion, an average of 9 weeks
  A full descriptive analysis of participant use of study clinician support will be conducted to assess scalability (CCBT-I arm only). This will be recorded through an electronic log by the study clinician following each contact with a participant. The unit of measure will include items such as the frequency of contact with the study clinician and a qualitative analysis of the nature of the support given.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Brenner, PhD, Principal Investigator — Rocky Mountain VA Mental Illness, Research, and Education Center
Locations (1):
- Rocky Mountain Regional VAMC, Aurora, Colorado, United States